CLINICAL TRIAL: NCT06602167
Title: Electroacupuncture Combined With Self-administered Acupressure for the Prevention of Capecitabine-Associated Hand-Foot Syndrome: a Randomized Controlled Trial
Brief Title: Electroacupuncture Combined With Self-administered Acupressure for the Prevention of Capecitabine-Associated Hand-Foot Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Jiuda Zhao, Clinical Professor, Affiliated Hospital of Qinghai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AHQU-2024001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Capecitabine; Hand-foot Syndrome; Electroacupuncture; Self-administered Acupressure; Breast Cancer; Gastrointestinal Cancers
Keywords: electroacupuncture; capecitabine; self-administered acupressure; Hand-foot syndrome; Breast cancer; Gastrointestinal cancers
MeSH Terms: conditions — Hand-Foot Syndrome; Breast Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True electroacupuncture + True self-administered acupressure plus doctor-prescribed treatment group (Experimental): True electroacupuncture: Participants will receive two electroacupuncture treatments within the first week of each treatment cycle. The acupuncturist inserts the needle into the point and manipulates the needle until the feeling of "deqi" is achieved and reported by the participant. The electrical stimulation will be administered at a sustained frequency of 2Hz for 30 minutes. True self-administered acupressure: In weeks 2 and 3 of each treatment cycle, participants performed true self-administered acupressure, pressing each acupoint with their thumb to achieve "deqi" for three minutes. Doctor-prescribed treatment: At the beginning of capecitabine, patients will be treated with doctor-recommended medications, including oral celecoxib, topical diclofenac, and other skin protectants.
  Interventions: Combination Product: True electroacupuncture + True self-administered acupressure; Drug: Doctor-prescribed treatment
- Sham electroacupuncture + sham self-administered acupressure plus doctor-prescribed treatment group (Sham Comparator): Sham electroacupuncture: The sham electroacupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive acupuncture treatment without electrical stimulation same the intervention group. And avoid "deqi" sensation. Sham self-administered acupressure: administered non-acupressure points 1 to 3cm away from the true acupressure points used in the experimental group and away from known meridians. The frequency, course duration, and overall treatment time will be the same as those in the true self-administered shiatsu group. The applied pressure does not cause a feeling of "deqi". Doctor-prescribed treatment: All the drugs used are the same as those in the experimental group.
  Interventions: Drug: Doctor-prescribed treatment; Combination Product: Sham electroacupuncture + Sham self-administered acupressure

INTERVENTIONS:
Combination Product: True electroacupuncture + True self-administered acupressure — True electroacupuncture: Participants will receive two electroacupuncture treatments within the first week of each treatment cycle. The acupuncturist inserts the needle into the point and manipulates the needle until the feeling of "deqi" is achieved and reported by the participant. The electrical stimulation will be administered at a sustained frequency of 2Hz for 30 minutes. True self-administered acupressure: In weeks 2 and 3 of each treatment cycle, participants performed true self-administered acupressure, pressing each acupoint with their thumb to achieve "deqi" for three minutes.
  Arms: True electroacupuncture + True self-administered acupressure plus doctor-prescribed treatment group
Drug: Doctor-prescribed treatment — Doctor-prescribed treatment: At the beginning of capecitabine, patients will be treated with doctor-recommended medications, including oral celecoxib, topical diclofenac, and other skin protectants.
Combination Product: Sham electroacupuncture + Sham self-administered acupressure — Sham electroacupuncture: The sham electroacupuncture comprised a core standardized prescription of minimally invasive, shallow needle insertion using thin and short needles at body locations not recognized as true acupuncture points and are deemed to not belong to traditional Chinese meridians and have no therapeutic value. Participants will receive acupuncture treatment without electrical stimulation same the intervention group. And avoid "deqi" sensation. Sham self-administered acupressure: Administered non-acupressure points 1 to 3cm away from the true acupressure points used in the experimental group and away from known meridians. The frequency, course duration, and overall treatment time will be the same as those in the true self-administered shiatsu group. The applied pressure does not cause a feeling of "deqi".
  Arms: Sham electroacupuncture + sham self-administered acupressure plus doctor-prescribed treatment group

SUMMARY:
This study hypothesizes that electroacupuncture combined with self-administered acupressure plus doctor-prescribed treatment is effective in preventing Hand-Foot Syndrome (HFS) caused by capecitabine. It aims to explore the effectiveness of this combined approach in preventing HFS in patients with malignant tumors undergoing oral capecitabine treatment. Further exploration of prevention and treatment methods may enhance the quality of life for patients during the treatment process.

DETAILED DESCRIPTION:
This study is a parallel-group, blinded (blinding applies to participants, evaluators, investigators, and statisticians) randomized controlled trial designed to explore the preventive effect of electroacupuncture combined with self-administered acupressure plus doctor-prescribed treatment on HFS in patients with malignant tumors receiving oral capecitabine and to improve the quality of life for patients during treatment. Participants are randomly assigned to one of two groups: a true electroacupuncture combined with true self-administered acupressure group, or a sham electroacupuncture combined with sham self-administered acupressure group. The true electroacupuncture combined with true self-administered acupressure group receives true electroacupuncture combined with true self-administered acupressure plus doctor-prescribed treatment(oral administration of celecoxib, external application of diclofenac, and other skin protectants). The sham electroacupuncture combined with sham self-administered acupressure group receives sham electroacupuncture combined with sham self-administered acupressure plus the same doctor-prescribed treatment. HFS will be assessed following the initiation of capecitabine treatment, with records kept of the capecitabine dosage, the severity of HFS, onset time, and duration of symptoms. In addition, the HFS-14 questionnaire was used to assess the condition of patients at each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form;
2. Male or female ≥ 18 years old;
3. Patients with gastrointestinal cancer or breast cancer who are diagnosed with cancer by pathology will receive capecitabine treatment for the first time according to the label;
4. The performance status of the Eastern Cancer Collaboration Group is 0-2;
5. Palliative or adjuvant chemotherapy with capecitabine (combination or monotherapy, minimum daily total dose of capecitabine 2000 mg/m^2);
6. Expected lifespan ≥ 3 months;
7. Laboratory requirements: platelet count ≥ 100 × 10^9/L, white blood cell count>3.0 × 10^9/L, hemoglobin ≥ 10.0 g/dL, normal liver and kidney function;
8. Adequate contraception.

Exclusion Criteria:

1. Previous use of capecitabine or liposome doxorubicin or any other tyrosine kinase inhibitor that may induce HFS (such as sorafenib, sunitinib, and apatinib) for chemotherapy;
2. The initial dose of capecitabine is less than 800mg/m^2;
3. Radiation therapy or surgery should be performed within 4 weeks before the start of treatment;
4. Skin diseases that may interfere with clinical trial results;
5. Known drug/alcohol abuse;
6. Pregnant women or lactating patients;
7. Participate in another clinical trial and the patient has received the investigational drug within the last 30 days prior to the start of treatment (i.e. follow-up in the previous trial was not exclusive);
8. Known patients who are afraid of electroacupuncture stimulation or allergic to stainless steel needles or any component of capecitabine;
9. Receive any acupuncture and moxibustion treatment ,there is lymphedema in the area stimulated by acupuncture;
10. Patients with any chemotherapy- or radiotherapy-related toxicities that have not subsided to grade 2 or lower will be excluded, except for stable sensory neuropathy.
11. Any unresolved skin toxicity caused by previous chemotherapy or radiotherapy, except for hair loss, will also be grounds for exclusion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
HFS incidence rate (Compare the difference between the two groups) | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 1: Minimal skin changes or dermatitis (eg, erythema, oedema, or hyperkeratosis) without pain； Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.

SECONDARY OUTCOMES:
The incidence of HFS grade 2-3 (Compare the difference between the two groups) | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; ; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.
The occurrence time of grade 1-3 HFS (Compare the difference between the two groups) | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 1: Minimal skin changes or dermatitis (eg, erythema, oedema, or hyperkeratosis) without pain； Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.
The occurrence time of grade 2-3 HFS (Compare the difference between the two groups) | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.
The difference in duration (weeks) of grade 1 to 3 HFS between the two groups | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 1: Minimal skin changes or dermatitis (eg, erythema, oedema, or hyperkeratosis) without pain； Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.
The difference in duration (weeks) of grade 2 to 3 HFS between the two groups | Capecitabine started treatment until 12 weeks after the end of treatment
  The clinician evaluated the patient's HFS grade according to the NCI CTCAEv5.0 grading for HFS.
  Grade 2: Skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting instrumental activities of daily living; Garde 3: Severe skin changes (eg, peeling, blisters, bleeding, oedema, or hyperkeratosis) with pain; limiting self-care activities of daily living.
  The more severe the grade, the more it affects the quality of life of patients.
The time when pain/sensory abnormalities occur (Compare the difference between the two groups) | Capecitabine started treatment until 12 weeks after the end of treatment
  The time when pain/sensory abnormalities occur
Correlation between capecitabine dose and HFS grade | Capecitabine started treatment until 12 weeks after the end of treatment
  The correlation between the dose of capecitabine used by the patient and the grade of HFS was recorded.
The dependence of electroacupuncture and self-acupoint acupressure treatment in experimental group and control group | Capecitabine started treatment until 12 weeks after the end of treatment
  Rate of adherence to electroacupuncture therapy in experimental and control groups
Changes in patient reported results and adverse events using the HSF-14 (Hand-Foot Syndrome-14) scale from baseline to the end of the study | From the beginning to the end of capecitabine treatment
  The HSF-14 (Hand-Foot Syndrome-14) scale is a tool used to evaluate the severity of symptoms and their impact on quality of life in patients with HFS. A total of 14 items are included. Each item was scored on a three-point Likert scale: 0, "no, never"; 1, "yes, from time to time"; 2, "yes, always." Two separate questions were also added, one to measure limb involvement (type of limb affected by HFS, one or both) and one to measure pain. The limb involvement item was scored either 1if only the hands or feet were affected or 3 if both the hands andfeet were affected. The pain item was scored on a three-point scale: 1, not painful; 2, moderately painful; 3, very painful. The total HFS-14 score was calculated by summing the scores of all items and was adjusted to 100 by applying a rule of three. HFS-14 scores were in the range of 2-100, with the higher the score, the greater the quality of life impairment. For details, see PMCID: PMC3228077.

CONTACTS AND LOCATIONS:
Locations (1):
- Qinghai University Affiliated Hospital, Xining, Qinghai, China